CLINICAL TRIAL: NCT07284628
Title: A Phase II Drug Repurposing Trial of Vortioxetine for the Treatment of Patients With Newly Diagnosed Glioblastoma
Brief Title: Vortioxetine for Newly Diagnosed Glioblastoma
Acronym: ReVoGlio
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other); University Hospital, Basel, Switzerland (Other); Cantonal Hospital of St. Gallen (Other); Kantonsspital Aarau (Other); Cantonal Hospital of Lucerne, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReVoGlio
Record Dates: First submitted 2025-09-28; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Drug repurposing; Vortioxetine
MeSH Terms: conditions — Glioblastoma | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortioxetine in addition to the standard of care (Experimental)
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine will be added to standard of care temozolomide chemoradiotherapy for patients with newly diagnosed glioblastoma

SUMMARY:
There is a very urgent need to improve on the currently limited treatment options for patients with glioblastoma. Despite extensive knowledge on the molecular pathogenesis of glioblastoma obtained through genomic, transcriptional and proteomic profiling, targeted therapy efforts have not yielded major advances, likely because of interindividual and intraindividual tumor heterogeneity and redundant oncogenic pathway activation.

Accordingly, there is a strong rationale to approach the challenge of glioblastoma from a different angle, e.g., by ex vivo drug sensitivity profiling which is agnostic to the molecular profile of a tumor. This approach that we have termed "pharmacoscopy", has previously been explored in liquid cancers and probably led to improved patient outcomes. Using pharmacoscopy, the antidepressant drug, vortioxetine, has been identified as a lead candidate for further exploration in patients with glioblastoma. Vortioxetine also demonstrated synergistic anti-glioma activity in combination with temozolomide or lomustine.

The ReVoGlio trial aims at demonstrating that vortioxetine, a drug selected based on ex vivo drug profiling (pharmacoscopy), is of benefit for patients with newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years
2. Patients with histologically confirmed newly diagnosed glioblastoma per CNS WHO 2021 classification
3. O6-methylguanine DNA methyltransferase (MGMT) promotor methylation status known or tissue available for testing
4. Karnofsky performance status (KPS) ≥ 70%
5. Intent to treat with standard radiochemotherapy per EANO guidelines (radiotherapy will 60 Gy in 1.8-2 Gy fractions. Concomitant chemotherapy with temozolomide (75 mg/m2 daily throughout radiotherapy, including at weekends) followed by six cycles of maintenance temozolomide (150-200 mg/m2, 5 out of 28 days). Short course radiotherapy at 40 Gy is not allowed.
6. Female patients must be either documented not to be Women of Childbearing Potential (WOCBP) or must have a negative pregnancy test within 14 days of starting treatment. Additionally WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner. WOCBP are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).
7. Male subjects able to father children must agree to use two acceptable methods of contraception throughout the study and during 6 months following the last study drug administration (e.g., condom with spermicidal gel). Double-barrier contraception is required.
8. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
9. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Prior treatment for newly diagnosed glioblastoma except surgery. 2. Intent to be treated with tumor-treating fields. 3. Inability to undergo contrast-enhanced MRI. 4. Inadequate bone marrow, renal and hepatic function:

* Absolute neutrophil count (ANC) < 1.5 x 10.9/L; platelets < 100 x 10.9/L
* Hemoglobin (Hb) < 9.0 g/dl. Blood marrow values must be measured independently of transfusion.
* Chronically impaired renal function as indicated by creatinine clearance < 50 mL/min or serum creatinine > 1.5 upper limit of normal (ULN).
* Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN) 9. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.

  10. Any contra-indication to vortioxetine. 11. Medically documented history of active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g., risk of doing harm to self or others), or patients with active severe personality disorders.

  12. Pregnancy or breast feeding. 13. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.

  14. Concurrent malignancies unless the patient has been disease-free without intervention for at least one year.

  15. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion for each patient, an average of 6 months
  PFS is defined as the time from registration until the first event of interest: progressive disease or death from any cause. Patients not having an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting a new treatment. The PFS will be determined locally per RANO 2.0 criteria

SECONDARY OUTCOMES:
Adverse events | From date of randomization until 30 days after vortioxetine interruption
  All AE will be assessed according to CTCAE v5.0
Overall survival (OS) | until death, an average of 17 months
  OS will be calculated from registration until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive. OS will be assessed in relation to external control data.
Neurological function 1 | through study completion for each patient, an average of 6 months
  measured by NANO scale
Neurological function 2 | through study completion for each patient, an average of 6 months
  measured by the RANO seizure scale
Neurological function 3 | through study completion for each patient, an average of 6 months
  measured by Karnofsky performance status
Neurological function 4 | through study completion for each patient, an average of 6 months
  measured by steroid consumption
Quality of life 1 | through study completion for each patient, an average of 6 months
  assessed by QLQ C30 questionnaire
Quality of life 2 | through study completion for each patient, an average of 6 months
  assessed by BN20 questionnaire
Anxiety | through study completion for each patient, an average of 6 months
  assessed by the Hamilton Anxiety Rating Scale (HAM-A) (Hamilton 1959)
Response to treatment | through study completion for each patient, an average of 6 months
  Response (type of response and response rate per local and central assessment in patients with measurable disease) and progression-free survival to treatment by central review of the MRI

OTHER OUTCOMES:
Prognostic role of extent of resection and residual tumor | until death, an average of 17 months
  Assessment of a statistical association between extent of surgical resection / residual tumor (measured in mm3) and outcome (survival)
Prognostic role of the G8 frailty index | through study completion for each patient, an average of 6 months
  Assessment of a statistical association between the G8 total score and outcome (survival)
Drug exposure | through study completion for each patient, an average of 6 months
  Plasmatic concentration of vortioxetine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Weiss T, Buhler M, Mena J, Lottenbach Z, Wegmann R, Sun M, Bihl M, Augustynek B, Baumann SP, Goetze S, van Drogen A, Pedrioli PGA, Penton D, Festl Y, Buck A, Kirschenbaum D, Zeitlberger AM, Neidert MC, Vasella F, Rushing EJ, Wollscheid B, Hediger MA, Weller M, Snijder B. High-throughput identification of repurposable neuroactive drugs with potent anti-glioblastoma activity. Nat Med. 2024 Nov;30(11):3196-3208. doi: 10.1038/s41591-024-03224-y. Epub 2024 Sep 20. PMID 39304781